CLINICAL TRIAL: NCT01752023
Title: A Randomized Phase II Study of SUBATM-itraconazole With Cisplatin/Gemcitabine in Patients With Previously Untreated Metastatic Squamous Non-Small Cell Lung Cancer.
Brief Title: A Randomized Phase II Study of SUBATM-itraconazole in Patients With Untreated Squamous NSCLC.
Acronym: NA_00067809
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1230; NA_00067809 (Other: JHMIRB)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin + Gemcitabine with SUBATM-itraconazole (Experimental): SUBATM-itraconazole 200 mg BID, Cisplatin 75 mg/m2 day 1, Gemcitabine 1000 mg/m2 days 1 + 8 for 6 cycles. Then SUBATM-itraconazole 200 mg BID alone.
  Interventions: Drug: Cisplatin + Gemcitabine with SUBATM-itraconazole
- Cisplatin + Gemcitabine (Active Comparator): Arm B = Cisplatin 75 mg/m2 day 1, Gemcitabine 1000 mg/m2 days 1 + 8 for 6 cycles. Then Best supportive care.
  Interventions: Drug: Cisplatin + Gemcitabine

INTERVENTIONS:
Drug: Cisplatin + Gemcitabine with SUBATM-itraconazole — Experimental Arm
  Other Names: SUBATM-itraconazole + Cisplatin and Gemcitabine for 6 cycles followed by SUBATM-itraconazole alone.
  Arms: Cisplatin + Gemcitabine with SUBATM-itraconazole
Drug: Cisplatin + Gemcitabine — Active Comparator
  Other Names: Cisplatin and Gemcitabine for 6 cyles followed by Best supportive care.
  Arms: Cisplatin + Gemcitabine

SUMMARY:
Response rates.

Changes in tumor blood flow.

DETAILED DESCRIPTION:
To determine the objective response rates of cisplatin and gemcitabine with or without SUBATM-itraconazole in patients with chemotherapy-naïve metastatic squamous non-small cell lung cancer.

To assess the changes in tumor blood flow as measured by contrast enhanced MRI scanning in patients with metastatic squamous non-small cell lung cancer treated with cisplatin and gemcitabine with or without SUBATM-itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV squamous cell lung cancer, with no prior systemic chemotherapy.
* Patients who have received prior adjuvant chemotherapy for early-stage lung cancer are eligible if at least 6 months have elapsed from completion of that treatment.
* Patients whose tumors contain mixed non-small cell histologies are eligible if squamous carcinoma is the predominant histology. Mixed tumors with small cell anaplastic elements are not eligible.
* Patient must have measurable disease per RECIST 1.1 (defined in section 9.1.2).
* Patients with previous radiotherapy as definitive therapy for locally advanced non-small cell lung cancer are eligible, as long as the recurrence is outside the original radiation therapy port. Radiation therapy must have been completed greater than or equal to 2 weeks prior to enroll in this study.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of itraconazole or SUBATM-itraconazole in combination with gemcitabine/cisplatin in patients under 18 years of age, such patients are excluded from this study. Squamous cell lung cancer is exceedingly rare in children.
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group performance status 0 - 1.
* Patients must have adequate organ and marrow function.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with gemcitabine, cisplatin (except in the adjuvant setting), itraconazole or SUBATM-itraconazole.
* Uncontrolled brain metastases. Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to itraconazole, SUBATM-itraconazole, gemcitabine, cisplatin or other agents used in the study.
* Itraconazole is a strong CYP3A4 inhibitor and may increase plasma concentrations of drugs metabolized by this pathway. Co-administration of cisapride, midazolam, pimozide, quinidine, lovastatin, simvastatin, triazolam, dofetilide, or levacetylmethadol (levomethadyl) with SUBATM-itraconazole or itraconazole is contraindicated.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because itraconazole is Class C agent and both gemcitabine and cisplatin are Class D agents, with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SUBATM-itraconazole and gemcitabine/cisplatin, breastfeeding should be discontinued if the mother is to be treated on this protocol.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SUBATM-itraconazole, gemcitabine, or cisplatin with these essential mediations.
* Medical contra-indication to MRI (e.g. gadolinium allergy, or severe claustrophobia).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ettinger, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Bayview Medical Center at Johns Hopkins, Baltimore, Maryland
  - Johns Hopkins University, SKCCC, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin + Gemcitabine With SUBATM-itraconazole: SUBATM-itraconazole 200 mg BID, Cisplatin 75 mg/m2 day 1, Gemcitabine 1000 mg/m2 days 1 + 8 for 6 cycles. Then SUBATM-itraconazole 200 mg BID alone.
  Arm A: Experimental Arm
- Cisplatin + Gemcitabine: Arm B = Cisplatin 75 mg/m2 day 1, Gemcitabine 1000 mg/m2 days 1 + 8 for 6 cycles. Then Best supportive care.
  Arm B: Active Comparator
Period: Overall Study
Arm/Group | Cisplatin + Gemcitabine With SUBATM-itraconazole | Cisplatin + Gemcitabine
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: SUBATM-itraconazole 200 mg BID, Cisplatin 75 mg/m2 day 1, Gemcitabine 1000 mg/m2 days 1 + 8 for 6 cycles. Then SUBATM-itraconazole 200 mg BID alone.
  Arm A: Experimental Arm
- Arm B: Arm B = Cisplatin 75 mg/m2 day 1, Gemcitabine 1000 mg/m2 days 1 + 8 for 6 cycles. Then Best supportive care.
  Arm B: Active Comparator
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 59 [52 to 66] | 67 [67 to 67] | 66 [52 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates
Description: Per response evaluation criteria in solid tumors criteria
Time Frame: 6 weeks
Population: Trial closed due to early stopping rule, patients were not analyzed as there were only 3 patients enrolled.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Tumor Blood Flow.
Description: To assess the changes in tumor blood flow as measured by contrast enhanced MRI scanning in patients with metastatic squamous non-small cell lung cancer treated with cisplatin and gemcitabine with or without SUBATM-itraconazole.
Time Frame: 6 weeks.
Population: Study closed due to early stopping rule. There were only 3 patients enrolled which were therefore not analyzed.
Arm/Group | Cisplatin + Gemcitabine With SUBATM-itraconazole | Cisplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Median Time to Progression
Description: To determine the median time to progression and median duration of survival of patients with metastatic squamous non-small cell lung cancer treated with cisplatin and gemcitabine with or without SUBATM-itraconazole.
Time Frame: 2 years.
Population: Study closed due to early stopping rule. There were only 3 patients enrolled which were therefore not analyzed.
Arm/Group | Cisplatin + Gemcitabine With SUBATM-itraconazole | Cisplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Effects
Description: To characterize the adverse effects of cisplatin and gemcitabine with or without SUBATM-itraconazole in this patient population.
Time Frame: 2 years.
Population: Study closed due to early stopping rule. There were only 3 patients enrolled which were therefore not analyzed.
Arm/Group | Cisplatin + Gemcitabine With SUBATM-itraconazole | Cisplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Itraconazole Exposure Parameters
Description: To correlate itraconazole exposure parameters with median time to progression and median survival in this patient population.
Time Frame: 2 years.
Population: Study closed due to early stopping rule. There were only 3 patients enrolled which were therefore not analyzed.
Arm/Group | Cisplatin + Gemcitabine With SUBATM-itraconazole | Cisplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Tumor Necrosis
Description: To assess changes in tumor necrosis in response to cisplatin and gemcitabine with or without SUBATM-itraconazole.
Time Frame: 2 years.
Population: Study closed due to early stopping rule. There were only 3 patients enrolled which were therefore not analyzed.
Arm/Group | Cisplatin + Gemcitabine With SUBATM-itraconazole | Cisplatin + Gemcitabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes